CLINICAL TRIAL: NCT03952234
Title: Phase-1, Dose Finding and Safety Study on L- Citrulline Treatment of Nitric Oxide Deficiency in MELAS
Brief Title: L-Citrulline Dose Finding Safety Study in MELAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of South Florida (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Fernando Scaglia, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-43576; U54NS078059 (NIH)
Record Dates: First submitted 2019-05-08; First posted 2019-05-16 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: MELAS Syndrome
Keywords: Mitochondrial; Encephalomyopathy; Metabolic strokes; Stroke-like episodes; Citrulline; Nitric Oxide
MeSH Terms: conditions — MELAS Syndrome | interventions — Citrulline

STUDY DESIGN:
Intervention Model Description: L-Citrulline
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose finding safety study (Other): In this study, the highest acceptable dose of an amino acid called citrulline will be established in people who have a mitochondrial disorder. Previous research conducted by several groups including our center at Baylor College of Medicine has determined that there is a deficiency of a compound called nitric oxide in people affected with MELAS.
  Interventions: Drug: L-Citrulline

INTERVENTIONS:
Drug: L-Citrulline — To determine the safest maximum dose of L-Citrulline which could be used as a potential treatment for adults with disorder of energy metabolism called MELAS
  Other Names: L-Citrulline powder

SUMMARY:
The main purpose of this study is to determine the safest maximum dose of an amino acid, citrulline, which will be used as potential treatment for adult patients with a disorder of energy metabolism called Mitochondrial Encephalomyopathy, Lactic Acidosis, and Stroke-like episodes (MELAS). Once established, this dose will be used in a future clinical trial.

DETAILED DESCRIPTION:
The human body is made of many cells and each cell contains many mitochondria. Mitochondria are called the powerhouses of the cell, because they produce the energy needed for a cell to be healthy and function the way it is meant to.

Diseases of the mitochondria affect the way the tissues and cells of the body make and use energy, and can affect almost all the different organs of the body like the brain and the muscles.

MELAS syndrome is one of the mitochondrial diseases; patients with this disease have different complications including stroke like episodes, headache, muscle weakness, fatigue, and hearing loss. One of the factors contributing to complications seen in patients with MELAS syndrome, in particular the stroke like episodes, is decreased amount of an element called nitric oxide. This element is made in the bodies from an amino acid called arginine. Amino acids are the building blocks of proteins. Proteins make the muscles in the bodies, and they are present in meat, chicken and fish.

In this study, the highest acceptable dose of an amino acid called citrulline will be established in participants who have a mitochondrial disorder. Previous research conducted by several groups including Baylor College of Medicine has determined that there is a deficiency of a compound called nitric oxide in patients affected with MELAS.

The lack of nitric oxide could cause constriction of blood vessels in the brain making it easier for these patients to have a metabolic stroke. The amino acid citrulline is a foundation for nitric oxide. In earlier studies, the investigator has found that there is more production of nitric oxide in the body when participants affected with MELAS take L-citrulline.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of MELAS (stroke-like events, seizures, exercise intolerance or muscle weakness).
2. Subject must be aged 18 to 65 years.
3. The m.3243A>G mutation in the MTTL1 gene.
4. Elevated plasma lactate (>2.2 mmol/L) taken at any point in the screening period (6 months prior to screening visit, including and up to the baseline visit).
5. Negative urine pregnancy test, if applicable.
6. Score of 26 or higher on the Montreal Cognitive Assessment (MOCA). -

Exclusion Criteria:

1. Evidence of acute illness or physical disability that may interfere with their ability to undergo the study.
2. Tobacco use
3. Orthostatic hypotension defined as a decrease in systolic blood pressure of 20 mm Hg, or a decrease in diastolic blood pressure of 10 mm Hg, between one and three minutes of standing when compared with blood pressure from the sitting or supine position at the baseline visit.
4. Presence of the following signs or symptoms in the past 12 months at grade 3 or higher based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03: hypotension, syncope, dizziness, blurred vision, fatigue, concentration impairment, nausea, vomiting, diarrhea, hypoglycemia, or headache.
5. > 2 seizures in week prior to baseline visit.
6. Hypotension defined as systolic blood pressure ≤ 90 mm Hg or diastolic blood pressure ≤ 60 mm Hg at the baseline visit.
7. Arginine supplementation within one week prior to baseline visit.
8. Inability to travel to the study site.
9. Subjects with no evidence of neurological disease, muscle weakness, or exercise intolerance.
10. Subjects with evidence of moderate to severe renal impairment ( eGFR < 60 mL/min/1.73 m2 ) at the baseline visit.
11. Subjects with poor cognitive ability to provide consent and to understand and report hypoglycemia.
12. Unwillingness of sexually active female subjects of childbearing age to practice reliable methods of contraception.
13. Intake of drugs that increase NO synthesis, vasodilators, or amino acid supplements that cannot be stopped during the study period.
14. Positive urine pregnancy test.
15. Score of less than 26 on the Montreal Cognitive Assessment (MOCA). -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Establishment of the maximum tolerable dose of L-citrulline in patients with MELAS syndrome by measuring the incidence of dose limiting toxicities (DLTs) | Eight weeks
  Measurement of the incidence of treatment-emergent adverse events in a safety and tolerability phase 1 study.
  The following Dose Limiting
  Toxicities (DLTs) will be measured:
  1. Treatment-related adverse events (AE) at grade 3 or higher, or worsening of baseline status, defined by increase of at least 2 grades, if baseline grade is ≤1. The AEs will be graded based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. Subjects will be specifically monitored for the occurrence of the following adverse events:
     1. Syncope
     2. Dizziness
     3. Blurred Vision
     4. Fatigue
     5. Concentration Impairment
     6. Nausea
     7. Vomiting
     8. Diarrhea
     9. Hypoglycemia
     10. Headache
  2. Orthostatic hypotension defined as a decrease in systolic blood pressure of 20 mm Hg, or a decrease in diastolic blood pressure of 10 mm Hg, within three minutes of standing when compared with blood pressure from the sitting or supine position.

SECONDARY OUTCOMES:
Changes in cerebral blood flow effected by the use of citrulline supplementation | Four weeks
  Changes in cerebral blood flow by using arterial spin-labeling (ASL) magnetic resonance imaging (MRI) will be measured in milliliters per 100 grams of tissue per minute at four weeks while on citrulline and compared to measurement at baseline in milliliters per 100 grams of tissue per minute before the use of citrulline
Changes in cerebrovascular reactivity effected by the use of citrulline supplementation | Four weeks
  Changes in cerebrovascular reactivity by using arterial spin-labeling (ASL) magnetic resonance imaging (MRI) will be measured in milliliters per 100 grams of tissue per minute at four weeks while on citrulline and compared to measurement in milliliters per 100 grams of tissue per minute at baseline before use of citrulline
Changes effected by the use of citrulline supplementation in the micromolar concentration of plasma amino acids citrulline, arginine, ornithine, and alanine levels. | Four weeks
  Concentrations of plasma citrulline, arginine, ornithine, and alanine will be measured at baseline before citrulline supplementation and at four weeks during citrulline supplementation to determine the changes in concentration in micromoles per liter
Changes effected by the use of citrulline in the micromolar concentration of plasma alanine and in the concentration of plasma lactate (expressed in millimole per liter) | Four weeks
  Concentrations of plasma lactate and plasma alanine will be measured at baseline before citrulline supplementation and at four weeks during citrulline supplementation to determine the change in concentration in micromoles per liter in plasma alanine and in millimoles per liter in plasma lactate
Changes effected by the use of citrulline in the concentration of plasma guanidino compounds | One week
  Concentration of plasma guanidino compounds will be measured at baseline before citrulline supplementation and at one week during citrulline supplementation by using untargeted metabolomics profiling and values will be expressed in Z scores

CONTACTS AND LOCATIONS:
Overall Officials: FERNANDO SCAGLIA, M.D, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor St. Luke'S Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Hattab AW, Emrick LT, Hsu JW, Chanprasert S, Almannai M, Craigen WJ, Jahoor F, Scaglia F. Impaired nitric oxide production in children with MELAS syndrome and the effect of arginine and citrulline supplementation. Mol Genet Metab. 2016 Apr;117(4):407-12. doi: 10.1016/j.ymgme.2016.01.010. Epub 2016 Jan 27. PMID 26851065
- [Background] El-Hattab AW, Almannai M, Scaglia F. MELAS. 2001 Feb 27 [updated 2018 Nov 29]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1233/ PMID 20301411
- [Background] El-Hattab AW, Almannai M, Scaglia F. Arginine and citrulline for the treatment of MELAS syndrome. J Inborn Errors Metab Screen. 2017 Jan;5:10.1177/2326409817697399. doi: 10.1177/2326409817697399. Epub 2017 Mar 24. PMID 28736735
- [Background] El-Hattab AW, Emrick LT, Williamson KC, Craigen WJ, Scaglia F. The effect of citrulline and arginine supplementation on lactic acidemia in MELAS syndrome. Meta Gene. 2013 Oct 15;1:8-14. doi: 10.1016/j.mgene.2013.09.001. eCollection 2013 Dec. PMID 25411654
- [Background] Scaglia F, Northrop JL. The mitochondrial myopathy encephalopathy, lactic acidosis with stroke-like episodes (MELAS) syndrome: a review of treatment options. CNS Drugs. 2006;20(6):443-64. doi: 10.2165/00023210-200620060-00002. PMID 16734497
- [Background] Hirano M, Pavlakis SG. Mitochondrial myopathy, encephalopathy, lactic acidosis, and strokelike episodes (MELAS): current concepts. J Child Neurol. 1994 Jan;9(1):4-13. doi: 10.1177/088307389400900102. PMID 8151079
- [Background] Noguchi T, Yoshiura T, Hiwatashi A, Togao O, Yamashita K, Nagao E, Shono T, Mizoguchi M, Nagata S, Sasaki T, Suzuki SO, Iwaki T, Kobayashi K, Mihara F, Honda H. Perfusion imaging of brain tumors using arterial spin-labeling: correlation with histopathologic vascular density. AJNR Am J Neuroradiol. 2008 Apr;29(4):688-93. doi: 10.3174/ajnr.A0903. Epub 2008 Jan 9. PMID 18184842
- See also: L-citrulline and Metformin in Duchenne's Muscular Dystrophy — https://clinicaltrials.gov/ct2/show/NCT01995032